CLINICAL TRIAL: NCT00738036
Title: Acute Pain Episodes in Patients Under Opioid Maintenance Therapy : Clinical Management and Long Term Effects
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 07 001 07
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Pain
Keywords: Analgesics; Opioid; Opioid maintenance therapy; Acute pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group P: Exposed to an acute painful phenomenon requiring an analgesic management
- Group C: Control, not exposed to acute pain

SUMMARY:
To define a rational pharmacological management of pain for the subjects under opioid maintenance therapy (methadone or buprenorphine), it is first of all necessary to estimate the efficiency of the current practices on pain management as well as their potentially noxious consequences, in particular on the long term opioid maintenance therapy.

The objective of the study is to compare the efficiency of the opioid maintenance therapy according to the arisen of an acute painful phenomenon requiring an analgesic management for these patients. At first, this work will allow to determine the results on acute pain of the current practices for these patients. The comparison of the long term consequences on opioid maintenance therapy between the patients that presented an acute painful phenomenon and the control patients should help to improve acute pain management for these patients while limiting the risk of relapse in the abused consumption of psychoactive substances.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more.
* Patients under opioid maintenance therapy (buprenorphine or methadone)
* Patients treated by the same drug (buprenorphine or methadone) since at least 3 months

Exclusion Criteria:

* Refusal of the patient to take part in the study
* Absence of possible follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under opioid maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Retention rate under buprenorphine or methadone treatment defined as the percentage of patients still under treatment during the follow-up | 1, 3, 6 and 12 months

SECONDARY OUTCOMES:
pain, anxiety, drugs, alcohol and other substances abuse and dependence, drug prescription (included for pain treatment and opioid maintenance) | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Lapeyre-Mestre, MD, Study Director — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Bounes V, Palmaro A, Lapeyre-Mestre M, Roussin A. Long-term consequences of acute pain for patients under methadone or buprenorphine maintenance treatment. Pain Physician. 2013 Nov-Dec;16(6):E739-47. PMID 24284855